CLINICAL TRIAL: NCT06790758
Title: Plasma Rich Fibrin Epidural Injection by Racz Catheter in Postdural Puncture Headache Guided Optic Nerve Sheath Diameter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR940/11/24
Record Dates: First submitted 2025-01-18; First posted 2025-01-24 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Plasma Rich Fibrin; Epidural; Racz Catheter; Postdural Puncture Headache; Optic Nerve Sheath Diameter
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plasma rich fibrin epidural injection by Racz catheter (Experimental): Patients will receive plasma-rich fibrin epidural injection by Racz catheter in post-dural puncture headache-guided optic nerve sheath diameter.
  Interventions: Drug: Plasma rich fibrin epidural injection by Racz catheter

INTERVENTIONS:
Drug: Plasma rich fibrin epidural injection by Racz catheter — Patients will receive plasma-rich fibrin epidural injection by Racz catheter in post-dural puncture headache-guided optic nerve sheath diameter.

SUMMARY:
This study aims to evaluate plasma-rich fibrin epidural injection by Racz catheter in post-dural puncture headaches guided optic nerve sheath diameter.

DETAILED DESCRIPTION:
Postdural puncture headaches (PDPHs) are a recognized complication following unintentional dural puncture during epidural analgesia or intentional dural puncture for spinal anesthesia, diagnostic, or interventional neuraxial procedures.

Plasma-rich fibrin (PRF) is derived from autologous whole blood that contains and releases several different growth factors and cytokines to stimulate the healing of bone and soft tissue via degranulation, which has recently gained popularity in pain management.

Optic nerve sheath diameter (ONSD) is important because the optic nerve is surrounded by subarachnoidal cerebrospinal fluid and all three meningeal layers, and a change in the ONSD can indicate changes in intracranial pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* Patients suffering from severe post-dural puncture headache.

Exclusion Criteria:

* Uncooperative patients.
* Severe comorbid conditions.
* Pregnancy.
* Anticoagulant therapy.
* Known allergies to plasma rich fibrin components.
* Body mass index (BMI) ≥35 kg/m2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-11-23 (Actual); Study Completion 2025-11-23 (Actual)

PRIMARY OUTCOMES:
Success rate of the procedure | 24 hours after the intervention
  Success rate plasma-rich fibrin for the treatment of headaches and associated symptoms on a 4-point rating scale (0 = none, 1 = slight, 2 = marked, 3 = complete relief) will be recorded.

SECONDARY OUTCOMES:
Degree of pain | 8 days postoperatively
  Degree of pain will be assessed using the Numeric Rating Scale (NRS). NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS will be assessed at (0, 6, 12, 24, 48) h, 3, 4, 5, 6, 7, 8 days postoperatively
Length of bed rest | 8 days postoperatively
  Length of bed rest after PRF and the efﬁcacy of plasma-rich fibrin for the treatment of headaches and associated symptoms on a 4-point rating scale (0 = none, 1 = slight, 2 = marked, 3 = complete relief) will be recorded.
Change in optic nerve sheath diameter | 6 hours after the procedure
  Change in optic nerve sheath diameter (ONSD) will be measured before and 6 hours after the procedure.
Incidence of complications | 8 days postoperatively
  Incidence of complications that may occur during the technique such as (bending of the tip of the needle, shearing of the catheter, misplacement of the catheter, blocking of the catheter, blood aspiration and bleeding in the epidural space, hypotension, migration of the catheter, paresthesia, headache and infection) will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.